CLINICAL TRIAL: NCT04051697
Title: The SEA-CHANGE Study: a Pilot Randomized Controlled Trial of the SElf-management After Cancer of the Head and Neck Group intErvention
Brief Title: The SEA CHANGE Study: A Self Management Intervention for Head and Neck Cancer Survivors
Acronym: SEA-CHANGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dublin City University (Other)
Collaborators: National University of Ireland, Maynooth (Other); Newcastle University (Other); St. James's Hospital, Ireland (Other); St. Luke's Hospital (Unknown); Royal Victoria Eye and Ear Hospital (Other Government)
Responsible Party: Principal Investigator, Pamela Gallagher, PhD, Prof Pamela Gallagher, Dublin City University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DIFA-2017-022; DIFA-2017-022 (Other Grant/Funding Number: Health Research Board)
Record Dates: First submitted 2019-07-22; First posted 2019-08-09 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer; Self-management; Intervention; Pilot Randomised Control Trial; Behavioural intervention; Quality of Life
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Two-armed (intervention vs usual care) non-blinded pilot randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care arm (No Intervention): Participants allocated to the control group will receive their usual care. Healthcare professionals within the designated sites will deliver aftercare treatment as usual, with no changes to the patient's clinical care. Participants in this arm do not receive the self-management intervention (SEA CHANGE).
- Intervention arm (Experimental): Participants in the intervention group will receive usual care and will be offered access to the self-management intervention (SEA CHANGE). Healthcare professionals within the designated sites will deliver aftercare treatment as usual, with no changes to the patient's clinical care.
  Interventions: Behavioral: SEA CHANGE intervention

INTERVENTIONS:
Behavioral: SEA CHANGE intervention — The SEA CHANGE intervention consists of six 2.5 hour facilitated group workshop sessions. The sessions run over six consecutive weeks and are delivered face-to-face by a leader and peer facilitator (HNC survivor). Each session focuses on a specific self-management topic and the development/enhancement of a particular set of skills. There are opportunities for peer learning, skills practice and take-home exercises to consolidate skills development. In delivering the intervention, leaders/facilitators use a standardised approach following a leader's/facilitators' manual and participant toolkit.
  Arms: Intervention arm

SUMMARY:
This study aims to test the feasibility of implementing the Self-Management after Cancer of the Head and Neck Group Intervention (SEA-CHANGE), designed to promote quality of life and participation in life activities and reduce distress in people who have completed primary treatment for head and neck cancer as compared to usual care.

DETAILED DESCRIPTION:
Head and neck cancer (HNC) and its treatment are associated with specific challenges such as facial disfigurement and impairments in speech, breathing and swallowing, and can have a negative impact on well-being. Self-management interventions can provide people with skills to deal with health-related problems, maintain life roles, and manage negative emotions, and have been found to increase confidence, improve quality of life, and reduce health service use across a range of chronic conditions.

The aim of this study is to pilot a self-management intervention (SEA-CHANGE) designed to promote quality of life and participation in life activities, and reduce distress in people who have completed primary treatment for HNC as compared to usual care. The study includes: (1) a pilot randomised study to assess the feasibility and acceptability of the intervention and its related procedures; (2) a qualitative process evaluation of the intervention; and (3) a systematic decision-making process regarding progression to a definitive trial. The expected outcome is a self-management intervention that is feasible and acceptable to HNC survivors and has the potential to realise both health benefits and economic gains.

ELIGIBILITY:
Inclusion Criteria:

* had a pathologically confirmed diagnosis of an invasive primary tumour in the head and neck (oral cavity, salivary glands, nasal cavity, sinuses, middle ear, pharynx and larynx);
* have undergone and completed treatment by surgery, chemotherapy, radiotherapy or a combination thereof;
* are aged 18 or older at the time of their HNC diagnosis;
* are within 12 months of having completed their primary treatment; and
* have provided written informed, consent.

Exclusion Criteria:

* are unable to read or speak English;
* had a second invasive primary cancer other than non-melanoma skin cancer diagnosed after the HNC (as these patients are likely to be more focused on the treatment of their second cancer rather than self-management of their HNC);
* are unable to provide informed consent (e.g., if they have dementia/Alzheimer's disease); or
* have other known medical condition or other reason why they would be unable to take part.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in the Functional Assessment of the Cancer Therapy scale (FACT-G and Head and Neck Cancer Subscale (FACT H&N)) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  FACT-G consists of 4 domains and 27 statements, asking participants to consider the previous week and rate their Quality of life (QoL) across physical, social/family, emotional, and functional domains on a five point likert scale (0-4). FACT H&N comprises 12 statements about HNC specific challenges and can be used independently of the FACT-G to indicate HNC specific QoL. Higher domain scores indicate higher QoL (Maximum domain scores: Physical 28; Social/Family 28; Emotional 24; Functional 28; FACT H&N subscale 48). The FACT-G and FACT H&N subscale have been widely used and validated and are commonly used to assess the QoL of HNC survivors.

SECONDARY OUTCOMES:
Changes in The Distress Thermometer scale from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The distress thermometer measures an individuals level of distress during the past week and is scored on a 0 to 10 point Likert scale with 0 indicating "No distress" and 10 indicating "Extreme distress". Scores of 4 or more indicate moderate to extreme distress.
Changes in the Social Role Participation Questionnaire (SRPQ) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The SRPQ assesses an individual's perceptions of: 1) the importance of participation in diverse roles; 2) restrictions in role participation; and 3) satisfaction with performance in social roles. Mean scores are calculated separately for each of the 3 social role dimensions on Likert scales: 1) salience or role importance (scores; 1 "Not at all important" to 5 "Extremely important"); 2) physical difficulty with each role (i.e., role limitations) (scoring; 1 "No difficulty" to 4 "Unable to do") and 3) satisfaction with role performance (scoring; 1 "Not satisfied" to 5 "Extremely satisfied"). Because individuals may not engage in all roles, mean role satisfaction scores are calculated if participants respond to at least 9 of 12 role domains.
Changes in the Fear of Recurrence/Relapse Scale from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The Fear of Recurrence/Relapse Scale is a five-item scale measuring patients' beliefs about recurrence of their cancer using 5-point Likert scales from 1 (Strongly agree) to 5 (Strongly disagree). Scores range from 5-25 and higher scores reflect a greater fear of cancer relapse.
Changes in the UK Cancer Costs Questionnaire (UKCC) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The UKCC is a modular questionnaire designed to capture the resources used by people with a current or previous diagnosis of cancer. Each question can be used in isolation. Captured activity includes primary care usage, community care usage, medications and personal social services. Societal costs are also captured including patient out-of-pocket costs, costs incurred by carers and time taken off work. The questionnaire has been appropriately modified for the Irish context.

OTHER OUTCOMES:
Changes in the Cancer Survivors' Self-efficacy Scale (CS-SES) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The CS-SES measures self-efficacy in cancer survivors' by assessing confidence in performing various disease-related activities. The scale consists of 11 items scored on a 10 point scale with 1 being "not at all confident" to 10 being "totally confident". An overall score is determined using the mean of the 11 items.
Changes in the Cognitive Emotional Regulation Questionnaire (CERQ) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The CERQ measures what an individual thinks after experiencing threatening or stressful life events using a 36 item questionnaire focused on 9 domains; self-blame, blaming others, rumination, catastrophizing, putting into perspective, positive refocusing, positive reappraisal, acceptance and planning. Each item is scored on a Likert scale ranging from 1 (Almost never) to 5 (Almost always). Individual sub-scales are calculated by summing the scores from individual sub-scales with a range from 4 to 20.
Changes in the Health Education Impact Questionnaire (HEIQ) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  The HEIQ is used as a measure of health education/ self-management behaviors in eight domains; Health Directed Behavior, Positive and Active Engagement in Life, Emotional Well-being, Self-monitoring and Insight, Constructive Attitudes and Approaches, Skills and Technique Acquisition, Social Integration and Support, and Health Service Navigation. Individuals are asked to indicate their level of agreement with 42 statements across the eight domains on four point Likert scales (1 "strongly disagree" to 4 "Strongly agree"). Higher scores indicate greater performance of specific self-management behaviors. Higher scores on the emotional well-being domain denote higher levels of negative affect. Each domain is used individually by calculating the mean score.
Changes in the Patient Activation Measure (PAM) from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  PAM assesses an individual's knowledge, skills and confidence for self-management. The measure contains 13 items measured on 4 point Likert scales (1 "Strongly disagree" to 4 "Strongly agree"). A total score is derived by dividing the raw score by the number of items answered and multiplying by 13. Calibration tables are used to apply a range of 1-100 with higher scores indicating higher patient activation.
Changes in lifestyle behaviours from baseline up to 12 months | 12 months; change from baseline (before randomisation) to post intervention, 6 months and 12 months
  Alcohol and tobacco use

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Gallagher, PhD, Principal Investigator — Dublin City University
Locations (3):
- Ireland (3):
  - Royal Victoria Eye and Ear Hospital, Ireland, Dublin
  - St James Hospital, Ireland, Dublin
  - St Lukes Hospital, Ireland, Dublin

IPD SHARING:
Plan to Share IPD: No